CLINICAL TRIAL: NCT02295033
Title: Phase III Study in the Conservative Management of Breast Carcinoma by Tumorectomy and Radiotherapy: Assessment of the Role of a Booster Dose of Radiotherapy (Joint Study of the European Organisation for Research and Treatment of Cancer Radiotherapy Cooperative Group and Breast Cancer Cooperative Group)
Brief Title: Randomized Boost Versus no Boost Irradiation of Early Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-22881-10882-ROG-BCG
Record Dates: First submitted 2014-11-17; First posted 2014-11-19 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Breast Cancer
Keywords: Boost versus no boost irradiation of early breast cancer
MeSH Terms: conditions — Breast Neoplasms

ARMS (2):
- Boost irradiation (Experimental)
  Interventions: Radiation: Boost irradiation
- No boost irradiation (No Intervention)

INTERVENTIONS:
Radiation: Boost irradiation
  Arms: Boost irradiation

SUMMARY:
Radiation therapy may kill any tumor cells remaining after surgery. This randomized phase III trial is studying the effect of an extra dose of radiation therapy (Boost dose) after breast conserving surgery and 50 Gy adjuvant external beam radiotherapy to see how well it works compared to no further therapy in treating women with early breast cancer that has been surgically removed.

DETAILED DESCRIPTION:
This is a randomized study. Patients are stratified by participating institution, menopausal status, clinical tumor size, nodal status, presence of Ductal Carcinoma In Situ, age, and resection margin status.

The objective of this trial is to assess the local recurrence rate and the cosmetic result in women who have had conservative resection of small breast cancers and who are randomly assigned after postoperative whole-breast irradiation to no boost vs. 15-16 Gy boost (patients with microscopically complete resections) or 10 Gy vs. 25-26 Gy boost (patients with microscopically incomplete resections).

Following tumorectomy, all patients receive radiotherapy for 5 weeks.

Patients with microscopically negative resection margins are randomized to one of 2 groups: no further radiotherapy; or a radiotherapy boost with either external-beam radiotherapy or an interstitial implant.

Patients with microscopically positive resection margins are also randomized to receive either lower dose or higher dose radiotherapy boosts by external beam or interstitial implant.

Patients with positive lymph nodes are encouraged to receive at least 6 courses of adjuvant or perioperative chemotherapy prior to radiotherapy provided radiotherapy is initiated within 6 months of surgery. All other patients begin radiotherapy within 9 weeks of surgery. All postmenopausal women with positive lymph nodes receive oral tamoxifen daily for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented invasive adenocarcinoma (any subtype) of the breast with clinical stage T1-2 (0-5 cm) and pathologic stage N0-1, M0 disease
* Lumpectomy with 1-2 cm margin required within 9 weeks of initiation of protocol radiotherapy
* Axillary dissection required for premenopausal patients and recommended for postmenopausal patients (Irradiation of clinically negative axilla is an acceptable alternative to axillary dissection in postmenopausal patients)

Exclusion Criteria:

* Residual microcalcification on postoperative mammogram
* Gross residual disease in the breast (re-excision allowed if there is gross residual disease after first surgical procedure)
* Multiple foci of tumor in more than 1 quadrant
* Previous or concurrent malignant tumor in contralateral breast
* In situ carcinoma of the breast, without invasive tumor
* Tumorectomy performed more than 9 weeks before the start of radiotherapy in cases where no adjuvant chemotherapy is given and more than 6 months before the start of radiotherapy if chemotherapy is given
* Previous history of malignant disease, except adequately treated carcinoma in situ of the cervix or basal cell carcinoma of the skin
* Concurrent pregnancy or lactation
* Eastern Cooperative Oncology Group performance scale more than 2

Max Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1989-05; Primary Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Time to local recurrence | 25 years from first patient in

REFERENCES:
- [Derived] Vrieling C, van Werkhoven E, Maingon P, Poortmans P, Weltens C, Fourquet A, Schinagl D, Oei B, Rodenhuis CC, Horiot JC, Struikmans H, Van Limbergen E, Kirova Y, Elkhuizen P, Bongartz R, Miralbell R, Morgan DA, Dubois JB, Remouchamps V, Mirimanoff RO, Hart G, Collette S, Collette L, Bartelink H; European Organisation for Research and Treatment of Cancer, Radiation Oncology and Breast Cancer Groups. Prognostic Factors for Local Control in Breast Cancer After Long-term Follow-up in the EORTC Boost vs No Boost Trial: A Randomized Clinical Trial. JAMA Oncol. 2017 Jan 1;3(1):42-48. doi: 10.1001/jamaoncol.2016.3031. PMID 27607734
- [Derived] Bartelink H, Maingon P, Poortmans P, Weltens C, Fourquet A, Jager J, Schinagl D, Oei B, Rodenhuis C, Horiot JC, Struikmans H, Van Limbergen E, Kirova Y, Elkhuizen P, Bongartz R, Miralbell R, Morgan D, Dubois JB, Remouchamps V, Mirimanoff RO, Collette S, Collette L; European Organisation for Research and Treatment of Cancer Radiation Oncology and Breast Cancer Groups. Whole-breast irradiation with or without a boost for patients treated with breast-conserving surgery for early breast cancer: 20-year follow-up of a randomised phase 3 trial. Lancet Oncol. 2015 Jan;16(1):47-56. doi: 10.1016/S1470-2045(14)71156-8. Epub 2014 Dec 9. PMID 25500422